CLINICAL TRIAL: NCT02355340
Title: Bone Mineral Density Status in Pediatric and Adolescent Survivors of Childhood Cancer With History of Bone Fracture
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Lynda Vrooman, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 14-411
Record Dates: First submitted 2015-01-23; First posted 2015-02-04 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Bone Mineral Density; Childhood Cancer Survivors
Keywords: Bone mineral density; Childhood cancer survivors
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DXA and pQCT Scan: * Dual energy x-ray absorptiometry (DXA): Assessment of bone mineral density
  * Peripheral quantitative computed tomography (pQCT): Assessment of bone mineral density
  Interventions: Other: Dual energy x-ray absorptiometry (DXA); Other: Peripheral quantitative computed tomography (pQCT)

INTERVENTIONS:
Other: Dual energy x-ray absorptiometry (DXA) — Subjects will undergo DXA scan to assess total body (less head) and lumbar spine bone mineral density.
Other: Peripheral quantitative computed tomography (pQCT) — Subjects will undergo pQCT assessment of radius and tibia.

SUMMARY:
This research study is evaluating bone mineral density in childhood cancer survivors who have a history of bone fracture.

DETAILED DESCRIPTION:
The purpose of this research study is to learn more about the status of bones in children and young-adults who have had bone fractures after treatment for childhood cancer. Bone complications including fracture can be important issues for some childhood cancer survivors. In this study we are measuring bone mineral density in children and young adults who have had bone fracture after treatment for childhood cancer. We will measure bone mineral density in two ways. We will use: 1) dual energy x-ray absorptiometry (also known as DXA), and 2) peripheral quantitative computed tomography (also known as pQCT).

ELIGIBILITY:
Inclusion Criteria:

* History of childhood cancer
* Age ≥ 8 years and < 20 years at time of enrollment
* ≥ 2 years since completion of cancer-directed therapy for first cancer
* Received chemotherapy for treatment of childhood cancer
* History of bone fracture after the conclusion of chemotherapy*
* Not currently receiving cancer-directed therapy
* Signed written informed consent (by parent if patient is < 18 years of age, or by patient, if he or she is ≥18 years of age)
* Patient assent for those ≥10 years of age and < 18 years of age for whom a parent provides informed consent (*History of bone fracture will be based on patient/parent report of fracture occurrence and will be confirmed in review of the medical record whenever feasible.)

Exclusion Criteria:

* Current treatment with bisphosphonates (as of time of enrollment)
* Current treatment with the anticonvulsant depakote (at time of enrollment)
* Currently pregnant

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood cancer survivors, currently age 8-20 with a history of bone fracture after completion of chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-05; Primary Completion 2024-06 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Total body BMD (total body less head) and lumbar spine BMD | Participants to undergo a single baseline assessment on day 1; to be measured at ≥ 2 years since completion of cancer-directed therapy
  DXA assessment (z-score)
Volumetric BMD of distal radius | Participants to undergo a single baseline assessment on day 1; to be measured at ≥ 2 years since completion of cancer-directed therapy
  pQCT assessment

SECONDARY OUTCOMES:
25-hydroxy vitamin D level | Participants to undergo a single baseline assessment on day 1; to be measured at ≥ 2 years since completion of cancer-directed therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Vrooman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts